CLINICAL TRIAL: NCT06468371
Title: Comparative Efficacy of Exercise Training Versus Dopamine Agonists in Treating Restless Legs Syndrome Among Hemodialysis Patients
Brief Title: Exercise Training Versus Ropinirole in Treating Restless Legs Syndrome Among Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Irfan Jamil, Dr., Lahore General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LahoreGeneralH
Record Dates: First submitted 2024-05-17; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Hemodialysis; Restless Legs Syndrome; ESRD (End Stage Renal Disease); Diabetes Complications
Keywords: ESRD (End Stage Renal Disease); Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome; Renal Insufficiency, Chronic; Diabetes Complications | interventions — Dopamine Agonists; ropinirole; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dopamine agonist (Active Comparator): * Ropinirole administration was begun with a dose of 0.25 mg, taken orally once daily, two hours before bedtime.
  * The dose was adjusted based on symptomatology at weekly intervals, with an increment of 0.5 mg, targeting a maximum dose of 2.0 mg, which was maintained for the remaining duration of the 12 weeks
  Interventions: Drug: Dopamine Agonist (Ropinirole)
- Excercise training (Experimental): * Exercise sessions involved using a pedal bicycle twice a week for 12 weeks, integrated into the patient's hemodialysis schedule.
  * Each exercise session lasted 20 minutes, scheduled between the second and third hours of dialysis.
  * The first 5 minutes were served as a warm-up, consisting of slow pedaling.
  * This was followed by 10 minutes of more intense pedaling.
  * After the initial 15 minutes, the pace was slow again for another 5 minutes for a cool-down period, helping to gradually reduce the heart rate.
  Interventions: Other: Excercise training

INTERVENTIONS:
Drug: Dopamine Agonist (Ropinirole) — Ropinirole administration will start at 0.25 mg orally once daily, two hours before bedtime. The dose will be adjusted weekly based on symptoms, increasing by 0.5 mg increments, up to a maximum of 2.0 mg, which will be maintained for the remaining 12 weeks.
  Other Names: Ropinirole
  Arms: Dopamine agonist
Other: Excercise training — Exercise sessions will involve using a pedal bicycle twice a week for 12 weeks, integrated into the patients' hemodialysis schedule. Each session will last 20 minutes, scheduled between the second and third hours of dialysis. The first 5 minutes will be for warm-up with slow pedaling, followed by 10 minutes of intense pedaling, and concluding with a 5-minute cool-down period of slow pedaling to gradually reduce the heart rate.
  Other Names: Physiotherapy
  Arms: Excercise training

SUMMARY:
This research aims to compare the efficacy of these two interventions, thereby addressing a critical gap in current therapeutic approaches. The rationale for this study is rooted in the existing evidence supporting non-pharmacological and pharmacological interventions for RLS, yet the comparative efficacy remains underexplored.

DETAILED DESCRIPTION:
The prevalence of end-stage kidney disease (ESKD) and its accompanying symptom burden, particularly restless legs syndrome (RLS), signified an urgent need for effective treatment strategies. RLS, with its higher prevalence in hemodialysis patients, posed significant challenges to their quality of life and overall health. Our hypothesis posited that there would be a significant difference in the effectiveness of exercise training versus dopamine agonist therapy in improving International Restless Legs Syndrome scores among hemodialysis patients. This research aimed to compare the efficacy of these two interventions, thereby addressing a critical gap in current therapeutic approaches. The rationale for this study was rooted in the existing evidence supporting non-pharmacological and pharmacological interventions for RLS, yet the comparative efficacy remained underexplored. The objective was to conduct a prospective comparative study within the Nephrology Department's Dialysis Unit at Sheikh Zayed Hospital, Rahim Yar Khan, with a sample size of 48, comprising 24 patients in each group. Adult patients, both male and female, diagnosed with ESKD and undergoing maintenance hemodialysis, who also met the criteria for RLS, were included. Group A received the dopamine agonist ropinirole, starting at a low dose (0.25 mg) and titrated according to symptomatology, while Group B underwent a structured exercise regimen on a pedal bicycle during their dialysis sessions. The outcome of this study was the change in IRLSS scores from baseline to 3 months post-intervention. Follow-up assessments were meticulously conducted to monitor these changes, with data recorded on a proforma designed for accuracy and consistency. Our data analysis plan involved chi-square or Fisher's exact test for categorical variables and independent t-tests for continuous variables, with a significance level set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18-60 years.
* Both male and female.
* Diagnosed with end-stage kidney disease (ESKD) and currently undergoing twice weekly maintenance hemodialysis for at least 3 months.
* Diagnosed with restless legs syndromeas defined by the International Restless Legs Syndrome Scale (IRLSS) criteria, with an IRLSSscore of 10 or higher at baseline.
* Able to participate in physical exercise as assessed by a healthcare professional.
* Patients must exhibit normal serum electrolyte levels, including potassium (3.5-5.0 mmol/L), calcium (8.5-10.2 mg/dL), phosphate (2.5-4.5 mg/dL), magnesium (1.7-2.2 mg/dL), and intact parathyroid hormone (iPTH) (150 to 600 pg/mL), as confirmed by recent laboratory tests.

Exclusion Criteria:

* Presence of other medical conditions that significantly impair mobility (e.g., severe arthritis, recent fractures, or amputations).
* Patients diagnosed with other neuropathies as assessed by neurologists.
* Patients in catabolic state with active infection, inflammation (C-reactive protein blood levels above 5.0 mg/l) or malignancy.
* Patients with diagnosed iron deficiency, defined by transferrin saturation less than 20%.
* Patients diagnosed with myocardial infarction or unstable angina over the last twelve months, existing heart failure or liver disease, poorly controlled diabetes (RBS ≥ 250 mg/dl) and uncontrolled hypertension with systolic blood pressure≥200 mmHg and /or diastolic blood pressure≥120 mmHg on two separate occasions.
* Patients requiring ≥13 mL/kg/hour ultrafiltration routinely as assessed by dialysis records.
* History of allergic reactions or contraindications to dopamine agonists if assigned to the pharmacological treatment group.
* Cognitive impairments or psychiatric conditions that may hinder understanding of the study requirements or compliance with the protocol.
* Patients refused to participate in the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in the International Restless Legs Syndrome Study Group (IRLSSG) score | From baseline to 3 months of interval.
  The IRLSS score is a validated instrument used to assess the severity of Restless Legs Syndrome (RLS). It comprises ten questions that evaluate the intensity of symptoms, their impact on sleep and daily life, and the frequency of symptom occurrence. Each question is rated on a scale from 0 (no symptoms) to 4 (severe symptoms). The overall score ranges from 0 to 40.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Irfan Jamil, MBBS, FCPS, Principal Investigator — Lahore General Hospital, Lahore
Locations (1):
- Lahore General Hospital, Lahore, Lahore, Punjab Province, Pakistan